CLINICAL TRIAL: NCT06143865
Title: Effects of Closed Aspiration on Hemodynamic Changes and Pain
Brief Title: Closed Aspiration on Hemodynamic Changes and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Elif Günay İsmailoğlu, Associate Professor, Izmir Bakircay University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BU-SBF-EI-002
Record Dates: First submitted 2023-07-05; First posted 2023-11-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Aspiration
Keywords: Closed aspiration; Pain; Hemodynamic parameters
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed aspiration group (Experimental): Closed system aspiration is performed according to standard guidelines for patients.
  Interventions: Procedure: Closed system aspiration

INTERVENTIONS:
Procedure: Closed system aspiration — Aspiration catheter; it is part of the ventilator and the ventilator circuit. The catheter is stored in a protective sheath. Therefore, the catheter can be used repeatedly during the day.

SUMMARY:
The study was planned to determine the effects of closed aspiration on arterial blood pressure, heart rate, respiratory rate, oxygen saturation level and pain in intensive care patients connected to mechanical ventilators. IThe effects of the closed aspiration system on hemodynamic parameters and pain will be determined and the results will be important in terms of the usability of the closed system in the clinical environment and raising awareness in nursing practices in order to create minimum complications for the patient.

DETAILED DESCRIPTION:
The research iss carried out in a single group pretest posttest quasi-experimental design in order to determine the effects of closed aspiration on arterial blood pressure, heart rate, respiratory rate, oxygen saturation level and pain in intensive care unit patients with mechanical ventilation. The research is carried out in Anesthesiology and Reanimation Intensive Care Unit. The sample of the study is patients who was intubated, not sedated, systolic arterial blood pressure 110-140 mmHg, diastolic arterial blood pressure between 60-90 mmHg, heart rate between 60-100/min, respiratory rate between 12-20/min, oxygen with saturation level (SpO2) >86%. Data is collected from the hospital's electronic patient record system and observationally before and after the aspiration. "Patient Description Form", "Hemodynamic Status and Pain Monitoring Form", "Behavioral Pain Scale" is used to collect research data.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years,
* Intubated
* Connected to mechanical ventilator,
* Not receiving sedation,
* Not unconscious,
* Monitored,
* Systolic arterial blood pressure is between 110-140 mmHg and diastolic arterial blood pressure is between 60-90 mmHg,
* Heart rate between 60-100/min,
* Respiratory rate between 12-20/min,
* Body temperature not higher than 38º C,
* Oxygen saturation level (SpO2) >86%

Exclusion Criteria:

* Not intubated,
* Received a diagnosis related to the respiratory system,
* Unconscious or sedated curare

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-07-10 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Hemodynamic status form 1 | 1 minute after aspiration.
  This form was used to record the arterial blood pressure, respiratory rate, oxygen saturation, heart rate of the patients.
Hemodynamic status form 2 | 5 minute after aspiration.
  This form was used to record the arterial blood pressure, respiratory rate, oxygen saturation, heart rate of the patients
Hemodynamic status form 3 | 30 minutes after aspiration.
  This form was used to record the hemodynamic parameters arterial blood pressure, respiratory rate, oxygen saturation, heart rate of the patients.
Behavioral pain scale 1 | 1st after aspiration.
  It consists of three items: facial expression, upper extremities, and compliance with the ventilator. For each item, there are four variables that include behavioral responses to pain. Each section is given a score between 1-4. The score obtained from the scale is between 3-12. Higher scores indicate increased pain intensity.
Behavioral pain scale 2 | 5th minutes after aspiration.
  It consists of three items: facial expression, upper extremities, and compliance with the ventilator. For each item, there are four variables that include behavioral responses to pain. Each section is given a score between 1-4. The score obtained from the scale is between 3-12. Higher scores indicate increased pain intensity.
Behavioral pain scale 3 | 30th minutes after aspiration.
  It consists of three items: facial expression, upper extremities, and compliance with the ventilator. For each item, there are four variables that include behavioral responses to pain. Each section is given a score between 1-4. The score obtained from the scale is between 3-12. Higher scores indicate increased pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Elif Günay İsmailoğlu, Izmir, Menemen, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No